CLINICAL TRIAL: NCT04733599
Title: High Frequency Spinal Cord Stimulation for Neuropathic Pain Following Brachial Plexus Avulsion Injury: a Prospective Observational Cohort Study
Brief Title: Neurostimulation for Treatment of Chronic Upper Limb Pain After Brachial Plexus Injury
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Christine (Christy) L. Hunt, Principal Investigator, Mayo Clinic
Other Study IDs: 20-000910
Record Dates: First submitted 2021-01-27; First posted 2021-02-02 (Actual); Last update posted 2025-05-26 (Actual); Status verified 2025-05

CONDITIONS: Brachial Plexus Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Adults with pain due to brachial plexus avulsion injury: Adult patients with history of brachial plexus avulsion injury referred for consideration of neuromodulation using high frequency neurostimulation will be considered.

SUMMARY:
The purpose of this study is to see how much pain intensity is affected by high frequency spinal cord stimulation therapy in individuals with serious brachial plexus injury.

DETAILED DESCRIPTION:
This single-site prospective observational cohort study will include all adults (> 18 years old) with brachial plexus avulsion injury who are candidates for high frequency (HF10) spinal cord stimulation (SCS). We plan to prospectively observe patients who undergo implantation of HF10 SCS for the indication of chronic neuropathic pain of the upper limb following brachial plexus avulsion injury.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Neuropathic pain of the upper limb ≥ 3 months following brachial plexus avulsion injury.
* Patients must be planned to undergo implantation of high-frequency spinal cord stimulation for the treatment of chronic neuropathic pain due to brachial plexus avulsion injury.

Exclusion Criteria:

* Pain that is non-neuropathic as defined by DN4 score <4.
* Pregnant at the time of consideration for implant or planning to become pregnant during the study duration.
* Active substance use disorder of any kind.
* Active tobacco use.
* Use of moderate or high dose opioid medication (oral morphine equivalents >100 mg daily).
* Active, untreated major psychiatric disorder that might interfere with subject's ability to participate.
* Involvement in active litigation related to injury.
* Patient has not undergone conservative medical management for at least 3 months (including physical and/or occupational therapy and at least one trial of neuropathic pain medication).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with history of brachial plexus avulsion injury referred to the Pain Clinic for consideration of neuromodulation using high frequency neurostimulation will be considered.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in neuropathic pain | Baseline, 1 month, 3 months, 6 months, 12 months, 18 months, 24 months, and 36 months
  Measured using the patient reported Neuropathic Pain Symptom Inventory (NPSI) which uses a scale of 0 = "have not felt such pain" and 10 = "feel it the worst" for a total score with a higher score indicates greater pain.
Change in multidimensional pain inventory | Baseline, 1 month, 3 months, 6 months, 12 months, 18 months, 24 months, and 36 months
  Measured using the West Haven-Yale Multidimensional pain inventory self-reported questionnaire to assess the impact of pain on daily living
Change in Douleur Neuropathique 4 (DN4) Questionnaire | baseline, 1 month, 3 months, 6 months, 12 months, 18 months, 24 months, and 36 months
  Change in DN4 questionnaire to estimate the probability of neuropathic pain with seven questions asking patients about quality of pain and three questions for physical examination of pain. Questions are yes = 1 or no = 0 to obtain a patient's total score out of 10, higher scores indicate more probability of pain.
Change in pain intensity | Baseline, 1 month, 3 months, 6 months, 12 months, 18 months, 24 months, and 36 months
  Measured using the PROMIS-CAT pain intensity scale
Change in pain interference | Baseline, 1 month, 3 months, 6 months, 12 months, 18 months, 24 months, and 36 months
  Measured using the PROMIS-CAT pain interference scale

SECONDARY OUTCOMES:
Change Disabilities of the Arm, Shoulder and Hand (DASH) disability/symptom score | Baseline, 1 month, 3 months, 6 months, 12 months, 18 months, 24 months, and 36 months
  Measured using the self-reported DASH 30-item questionnaire to assess the ability to perform activities. Total score on a scale of 0 indicating no disability to 100 indicating most serve disability
Assessment of the effectiveness of high frequency spinal cord stimulation in the above population in the improvement of quality of life as measured by validated patient-completed questionnaires. | baseline, 1 month, 3 months, 6 months, 12 months, 18 months, 24 months, and 36 months
  Measured using the EQ-5D.
Change in mood | Baseline, 1 month, 3 months, 6 months, 12 months, 18 months, 24 months, and 36 months
  Measured using the Center for Epidemiologic Depression Studies - Depression Scale. A 20-item self-reported questionnaire using a scale of 0 (rarely or none of the time) and 3 (most or all of the time) for a total score with high scores indicating the presence of more
Change in pain experience | Baseline, 1 month, 3 months, 6 months, 12 months, 18 months, 24 months, and 36 months
  Change in self-reported 13-item Pain Catastrophizing scale of 0 (not at all) and 4 (all the time) for a total score with higher scores indicating higher levels of pain anxiety
Change in pain anxiety | Baseline, 1 month, 3 months, 6 months, 12 months, 18 months, 24 months, and 36 months
  Measured using the self-reported Pain Anxiety Symptom Scale Short Form 20 to rate frequency of symptoms on a scale of 0 (never) to 5 (always) for a total score with higher score indicating high levels of pain-related anxiety
Assessment of the effect of high frequency spinal cord stimulation in the above population on sensory function in the affected limb. | Baseline, 1 month, 3 months, 6 months, 12 months, 18 months, 24 months, and 36 months
  Measured using Quantitative Sensory Testing

CONTACTS AND LOCATIONS:
Overall Officials: Christy Hunt, DO, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials